CLINICAL TRIAL: NCT02355522
Title: Randomized Controlled Trial of Local Lidocaine Gel and Intrauterine Lidocaine Infusion for Pain Relief During Saline Infusion Sonohysterography
Brief Title: Trial of Local Lidocaine Gel and Intrauterine Lidocaine Infusion for Pain Relief During Saline Infusion Sonohysterography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. YUNG Shuk Fei Sofie, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UW 13-294
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: saline infusion sonohysterography
MeSH Terms: conditions — Pain | interventions — K-Y jelly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lidocaine gel group (Active Comparator): 3ml of 2% lidocaine gel on the cervix and 5ml of intrauterine normal saline
  Interventions: Drug: Lidocaine gel; Drug: Intrauterine normal saline
- Intrauterine lidocaine group (Active Comparator): 3ml of KY jelly on the cervix and 5ml of 2% intrauterine lidocaine
  Interventions: Drug: Intrauterine lidocaine; Drug: KY jelly
- Placebo group (Placebo Comparator): 3ml of KY jelly on the cervix and 5mL of intrauterine normal saline
  Interventions: Drug: KY jelly; Drug: Intrauterine normal saline

INTERVENTIONS:
Drug: Intrauterine lidocaine
  Arms: Intrauterine lidocaine group
Drug: Lidocaine gel
  Arms: Lidocaine gel group
Drug: KY jelly
  Arms: Intrauterine lidocaine group; Placebo group
Drug: Intrauterine normal saline
  Arms: Lidocaine gel group; Placebo group

SUMMARY:
This is a randomized, double-blinded, double placebo-controlled trial. Patients undergoing saline infusion sonohysterography (SIS) will be recruited and randomized into three groups to receive (a) 3ml of 2% lidocaine gel on the cervix and 5ml of intrauterine normal saline; (b) 3ml of KY jelly on the cervix and 5ml of 2% intrauterine lidocaine or (c) 3ml of KY jelly on the cervix and 5mL of intrauterine normal saline prior to SIS. Pain levels will be recorded to evaluate the efficacy of local lidocaine gel and intrauterine lidocaine infusion in reducing pain during the SIS.

DETAILED DESCRIPTION:
Trial objectives and purpose:

To evaluate the efficacy of local lidocaine gel and intrauterine lidocaine infusion in reducing pain during saline infusion sonohysterography (SIS).

Trial design:

This is a randomized, double-blinded, double placebo-controlled trial. Patients undergoing SIS will be recruited and randomized into three groups to receive (a) 3ml of 2% lidocaine gel on the cervix and 5ml of intrauterine normal saline; (b) 3ml of KY jelly on the cervix and 5ml of 2% intrauterine lidocaine or (c) 3ml of KY jelly on the cervix and 5mL of intrauterine normal saline prior to SIS.

Randomization Before the procedure, each patient will be randomized into three groups with a predetermined computer-generated randomization code prepared by a research nurse to receive (a) 3ml of 2% lidocaine gel on the cervix and 5ml of intrauterine normal saline; (b) 3ml of KY jelly on the cervix and 5ml of 2% intrauterine lidocaine or (c) 3ml of KY jelly on the cervix and 5mL of intrauterine normal saline prior to SIS. Demographic data will be collected from all patients.

Blinding The test gel (2% lidocaine gel) and KY jelly are both colourless. They will be prepared by the research nurse and will not be labeled.

The study syringes containing test solution (lidocaine or normal saline) will also be prepared by the research nurse. Lidocaine and normal saline are identical in appearance (i.e., a clear colourless solution) and will be contained in identical 5-mL disposable syringes with labeled with numbers only.

The patient and the physician will not know the group allocation and what test gel and test solution are given. Only the research nurse responsible for the preparation knows about what the gel/solution are, but she will not be involved in the patient care, the procedure and the assessment of pain levels.

The procedure

Before the SIS, a sterile bivalve speculum will be introduced into the vagina for visualization of the cervix. The cervix and vagina will be cleansed with antiseptic solution. 3mL of test gel (2% lidocaine gel or KY jelly) will be applied to the surface of the cervix using a gauze according to group allocation. An infant feeding tube will be inserted into the uterine cavity through the endocervical canal. Test solution (2% lidocaine 5mL or normal saline 5mL) will be instilled into the uterine cavity through an infant feeding tube according to group allocation:

A) Lidocaine gel group: the subjects will receive local application of 2% lidocaine gel 3mL to the cervix (study drug) and intrauterine infusion of normal saline 5mL (placebo).

B) Intrauterine lidocaine group: the subjects will receive local application of KY jelly 3mL to the cervix (placebo) and intrauterine infusion of 2% lidocaine 5mL (study drug).

C) Placebo group: the subjects will receive local application of KY jelly 3mL to the cervix and intrauterine infusion of normal saline 5mL (double placebo).

The speculum will then be removed. After five minutes, the transvaginal ultrasound probe will be inserted into the vagina and 5 to 10 mL of sterile saline solution will be instilled into the uterine cavity. The volume of normal saline used depends on the distension of the uterine cavity, which should provide a clear visualization of the uterine cavity. After ultrasound examination, the transvaginal probe and the infant feeding tube will be removed, and the procedure is completed.

Assessment of pain levels

Patients will be asked to rate their pain levels during and after the procedure on a visual analogue scale (VAS), marking an "X" on a 10-cm line (0cm: no pain, 10cm: unbearable pain). Ratings will be done at different times:

1. just after speculum insertion
2. just after test solution (lidocaine or placebo) instillation
3. during normal saline infusion
4. immediately after the procedure
5. 20 minutes after the procedure
6. Overall pain score throughout the procedure The physician will also record and score visible signs of the women's distress during the procedure (moaning, body movement, grabbing the table, expressing about pain) using a 3-point observer scale for each of the parameters in which 0 is no response, 1 is mild response, and 2 is severe response. If the patient require additional analgesics, oral mefenamic acid 500 mg would be given and will be recorded.

Data collection Apart from assessment of pain levels, we will also record patient characteristics including age, parity, ethnicity, history of chronic pelvic pain, history of dysmenorrhea, prior curettage, menopausal status, education, socioeconomic status, indication of SIS, use of tenaculum, volume of saline solution infusion and presence of uterine pathologies. Any need for additional analgesics and side effects experienced by the subjects will be recorded. Blood pressure and pulse will be measured and recorded before and after the procedure.

Follow-up No routine follow-up visits will be arranged solely for the study unless considered necessary by the investigator.

Assessment of outcomes:

The primary outcome is the pain level during the SIS procedure as assessed by the visual analog scale. Other outcome measures include the patients' distress during, immediately and after the procedure as evaluated by the physician with a 3-point observer scale, the need for additional analgesics and side effects experienced by the patients.

Assessment of safety:

SIS is a well-established procedure to detect abnormalities of the uterus and endometrial cavity. It is a very safe procedure. It may cause cramping, spotting and vaginal discharge. Some women may experience severe pain and cramping. Pelvic infection occurs in less than 1%.

Lidocaine is a commonly used anaesthetic agent. Local application to the cervix and intrauterine use of lidocaine during various gynaecological procedures have been evaluated in several studies and no severe side effects were reported.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older being scheduled for saline infusion sonohysterography

Exclusion Criteria:

* History of cervical stenosis
* Known allergy to lidocaine
* Pregnancy
* Acute cervicitis
* Profuse vaginal bleeding
* Consumption of pain killers on the day of procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain level as assessed by the visual analog scale | Up to 20 minutues after the procedure
  Pain level during and after the saline infusion sonohysterography procedure as assessed by the visual analog scale

SECONDARY OUTCOMES:
Distress as evaluated by the physician with a 3-point observer scale | Just after the procedure
  Patients' distress during, immediately and after the procedure as evaluated by the physician with a 3-point observer scale
Analgesics | 1 hour
  Need for additional analgesics
Side effects | 1 hour
  Side effects experienced by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Sofie SF Yung, MBBS, MRCOG, FHKAM(O&G), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, China